CLINICAL TRIAL: NCT00713245
Title: A Long Term Follow up Study in Late-onset Pompe Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 200804012R
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Pompe Disease
Keywords: Pompe disease; late onset
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to observe the progression of disease in late-onset Pompe disease

ELIGIBILITY:
Inclusion Criteria:

* individuals with acid alpha glucosidase deficiency without obvious symptoms
* parents signed inform consent

Exclusion Criteria:

* individuals with acid alpha glucosidase deficiency presenting symptoms

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: individuals with acid alpha glucosidase deficiency but without obvious symptoms
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2008-05; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
all muscle function | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Whu-Liang Hwu, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan